CLINICAL TRIAL: NCT05070845
Title: AN INTERVENTIONAL PHASE 2, OPEN-LABEL, MULTI-CENTER STUDY TO EVALUATE SAFETY AND EFFICACY OF PF-06835375 IN ADULT PARTICIPANTS WITH MODERATE TO SEVERE PRIMARY IMMUNE THROMBOCYTOPENIA
Brief Title: Safety and Efficacy Study of PF-06835375 in Primary Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1131003; 2023-509338-21-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: ITP; platelets
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Open Label PF-06835375 dose 1 Treatment (Experimental): subcutaneous injection once monthly for 3 months
  Interventions: Biological: PF-06835375
- Open Label PF-06835375 dose 2 Treatment (Experimental): subcutaneous injection once monthly for 4 months
  Interventions: Biological: PF-06835375
- Open Label PF-06835375 dose 3 Treatment (Experimental): subcutaneous injection once monthly for 4 months
  Interventions: Biological: PF-06835375

INTERVENTIONS:
Biological: PF-06835375 — CXCR5 inhibitor

SUMMARY:
This is a Phase 2, open-label, multicenter, multiple subcutaneous injection, safety and efficacy study of PF-06835375 in adult participants with primary immune thrombocytopenia (ITP). This study will focus on participants with persistent (>3 months and ≤12 months), or chronic (>12 months) ITP

DETAILED DESCRIPTION:
This study is designed to elucidate the effects of PF-06835375 on platelet counts in participants with moderate to severe primary ITP. Based on the experience with other B-cells depleting agents, it is expected that the platelet counts will increase following a standard treatment. Each participant in cohort 1 will receive 1 subcutaneous injection of dose 1 every month for 3 months during the 12-week treatment period. And each participant in cohorts 2 and 3 will receive 1 subcutaneous injection of dose 2 or 3 every month for 4 months during the 16-week treatment period. This should provide sufficient levels of exposure and depletion of CXCR5 positive cells to sustain the effects of PF-06835375 during the treatment period. Additional depletion of Tfh cells may provide sustained increase in platelet count following the last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary ITP. Ongoing ITP (platelet counts <50 x 109/L) [No severe bleeding within 1 month or during screening] AND Persistent ITP (3 to 12 months) or Chronic ITP >12 months

Exclusion Criteria:

* Bleeding event according to the WHO grading scale ≥2 occurring ≤4 weeks prior to screen OR a current bleeding event that, in the opinion of the investigator, requires treatment with standard of care therapy OR require blood or blood products during screening
* Splenectomy within 3 months of randomization or planned during the study duration.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with change from baseline of platelet counts | baseline through 12 and 16 weeks
  To evaluate absolute value of platelet count of treated participants

SECONDARY OUTCOMES:
proportion of participants with modified overall response (mOR) | baseline through 12 and 16 weeks
  To evaluate the modified overall response of platelet count of treated participants
proportion of participants with complete response (CR) | baseline through 12 and 16 weeks
  To evaluate the complete response of platelet count of treated participants
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | baseline through end of study (Week 20 for cohort 1 and Week 24 for cohorts 2 and 3)
Proportion of participants with change from baseline of platelet counts | baseline to Week 20 and Week 24
Proportion of participants with change from baseline of circulating B cells | baseline to Week 20 and Week 24
Proportion of participants with change from baseline of circulating cTfh cells | baseline to Week 20 and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- East Carolina University, Greenville, North Carolina, United States
- Australia (9):
  - Clinical Research Unit Haematology, Division of Cancer Services, St. George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - South West Radiology, Liverpool, New South Wales
  - Slade Pharmacy, Mount Kuring-Gai, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - ICON Cancer Centre - Kurralta Park, Kurralta Park, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Canada (2):
  - Unity Health Toronto, St. Michael's Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Vseobecna fakultni nemocnice v Praze, Prague
- Hungary (4):
  - Pécsi Tudományegyetem Klinikai Központ, Pécs, Baranya
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County
  - Semmelweis University, Budapest
  - Petz Aladár Egyetemi Oktató Kórház, Győr
- Poland (6):
  - AIDPORT Sp. z o.o., Skórzewo, Greater Poland Voivodeship
  - InterHem, Bialystok
  - Klinika Hematologii i Transplantologii Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- United Kingdom (4):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Derriford Hospital, Plymouth, Devon
  - The Royal Cornwall Hospital, Truro, England
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1131003